CLINICAL TRIAL: NCT01752491
Title: A Phase I Trial of High-Dose Ascorbate in Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joseph J. Cullen, MD, FACS (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John M. Buatti, Professor and Chair, Department of Radiation Oncology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201211713; P30CA086862 (NIH); U01CA140206 (NIH)
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Glioblastoma; GBM; Glioblastoma Multiforme
Keywords: Ascorbate; Ascorbic acid; Vitamin C; Radiation; Temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — Ascorbic Acid; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 15g Ascorbate (Experimental): During radiation therapy:
  * Radiation: 61.2 Gray (1.8 Gray / fraction / day), 5 days/week, for approximately 8 weeks.
  * Temozolomide: 75 mg/m2, taken orally, once daily, every day, until radiation is completed.
  * Ascorbate: 15 g administered by IV three times a week until 1 month after radiation is completed (approximately 12 weeks).
  After radiation therapy:
  * Temozolomide: Starting 1 month after radiation. 150 mg/m2 and then 200 mg/m2 daily. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  * Ascorbate: escalating weekly doses of ascorbate (up to 125 grams) to target a serum level of 350 mg/dL (20 mM). Ascorbate is administered twice weekly, each week, for up to 6 months.
  Interventions: Drug: Ascorbate; Drug: Temozolomide; Radiation: Radiation therapy
- 25g Ascorbate (Experimental): If the 15g arm is tolerated, the study opens the 25g arm.
  During radiation therapy:
  * Radiation: 61.2 Gray (1.8 Gy/fraction/day), 5 days/wk, for about 8 weeks.
  * Temozolomide: 75 mg/m2, taken orally, once every day, until radiation is completed.
  * Ascorbate: 25 g administered by IV three times/wk until 1 month after radiation is completed (about 12 weeks).
  After radiation therapy:
  * Temozolomide: Starting 1 month after radiation. 150 mg/m2 and then 200 mg/m2 daily. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  * Ascorbate: escalating weekly doses of ascorbate (up to 125 grams) to target a serum level of 350 mg/dL (20 mM). Ascorbate is administered twice weekly, each week, for up to 6 months.
  Interventions: Drug: Ascorbate; Drug: Temozolomide; Radiation: Radiation therapy
- 50g arm (Experimental): If the 25g arm is tolerated, the study opens the 50g arm.
  During radiation therapy:
  * Radiation: 61.2 Gray (1.8 Gy/fraction/day), 5 days/wk, for about 8 weeks.
  * Temozolomide: 75 mg/m2, taken orally, once every day, until radiation is completed.
  * Ascorbate: 50 g administered by IV three times a week until 1 month after radiation is completed (about 12 weeks).
  After radiation therapy:
  * Temozolomide: Starting 1 month after radiation. 150 mg/m2 and then 200 mg/m2 daily. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  * Ascorbate: escalating weekly doses of ascorbate (up to 125 grams) to target a serum level of 350 mg/dL (20 mM). Ascorbate is administered twice weekly, each week, for up to 6 months.
  Interventions: Drug: Ascorbate; Drug: Temozolomide; Radiation: Radiation therapy
- 62.5g (Experimental): If the 50g arm is tolerated, the study opens the 62.5g arm.
  During radiation therapy:
  * Radiation: 61.2 Gray (1.8 Gy/fraction/day), 5 days/wk, for about 8 weeks.
  * Temozolomide: 75 mg/m2, taken orally, once every day, until radiation is completed.
  * Ascorbate: 62.5 g administered by IV three times a week until 1 month after radiation is completed (about 12 weeks).
  After radiation therapy:
  * Temozolomide: Starting 1 month after radiation. 150 mg/m2 and then 200 mg/m2 daily. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  * Ascorbate: escalating weekly doses of ascorbate (up to 125 grams) to target a serum level of 350 mg/dL (20 mM). Ascorbate is administered twice weekly, each week, for up to 6 months.
  Interventions: Drug: Ascorbate; Drug: Temozolomide; Radiation: Radiation therapy
- 75g Ascorbate (Experimental): If the 62.5g arm is tolerated, the study opens the 75g arm.
  During radiation therapy:
  * Radiation: 61.2 Gray (1.8 Gy/fraction/day), 5 days/wk, for about 8 weeks.
  * Temozolomide: 75 mg/m2, taken orally, once every day, until radiation is completed.
  * Ascorbate: 75 g administered by IV three times a week until 1 month after radiation is completed (about 12 weeks).
  After radiation therapy:
  * Temozolomide: Starting 1 month after radiation. 150 mg/m2 and then 200 mg/m2 daily. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  * Ascorbate: escalating weekly doses of ascorbate (up to 125 grams) to target a serum level of 350 mg/dL (20 mM). Ascorbate is administered twice weekly, each week, for up to 6 months.
  Interventions: Drug: Ascorbate; Drug: Temozolomide; Radiation: Radiation therapy
- 87.5g Ascorbate (Experimental): If the 75g arm is tolerated, the study opens the 87.5g arm.
  During radiation therapy:
  * Radiation: 61.2 Gray (1.8 Gy/fraction/day), 5 days/wk, for about 8 weeks.
  * Temozolomide: 75 mg/m2, taken orally, once every day, until radiation is completed.
  * Ascorbate: 87.5 g administered by IV three times a week until 1 month after radiation is completed (about 12 weeks).
  After radiation therapy:
  * Temozolomide: Starting 1 month after radiation. 150 mg/m2 and then 200 mg/m2 daily. Starting 28 days after the completion of radiation therapy. Taken for 5 days followed by 23 days of rest for 6 cycles.
  * Ascorbate: escalating weekly doses of ascorbate (up to 125 grams) to target a serum level of 350 mg/dL (20 mM). Ascorbate is administered twice weekly, each week, for up to 6 months.
  Interventions: Drug: Ascorbate; Drug: Temozolomide; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Ascorbate — Intravenous infusion of high-dose ascorbate
  Other Names: Ascorbic Acid; Vitamin C
Drug: Temozolomide — Oral chemotherapeutic
  Other Names: Temodar
Radiation: Radiation therapy — External beam radiation therapy
  Other Names: External beam radiation therapy

SUMMARY:
This is a phase 1 (first in man) study testing the safety of adding high dose ascorbate (vitamin C) to standard radiation and chemotherapy for initial treatment of glioblastoma multiforme (GBM).

DETAILED DESCRIPTION:
This phase 1 study will test the safety of adding high dose ascorbate (vitamin C) to standard chemoradiation and, after the radiation is completed, during 6 cycles of temozolomide.

Standard treatment for glioblastoma multiforme (GBM) involves surgery followed by radiation combined with temozolomide (a chemotherapy). After radiation, patients receive cycles of temozolomide (adjuvant chemotherapy)

Participants will:

* receive high doses of intravenous (IV) ascorbate three times a week during chemoradiation
* receive high doses of intravenous (IV) ascorbate twice a week during adjuvant chemotherapy (after radiation)

This is a phase 1 study will evaluate the side effects of adding this drug to the standard therapy. The dose given to a participant will be determined by how well other participants have tolerated the drug.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed (i.e., within 5 weeks), histologically or cytologically confirmed glioblastoma multiforme.
* Diagnosis must be made by surgical biopsy or excision.
* Therapy must begin ≤ 5 weeks after surgery.
* Age ≥ 18 years
* ECOG performance status 0-2 (Karnofsky > 50%).
* A complete blood count and differential must be obtained within 21 days prior to the first dose of radiation, with adequate bone marrow functions as defined below:

  * Absolute neutrophil count (ANC) ≥ 1500 cells per mm3
  * Platelets ≥ 100,000 per mm3
  * Hemoglobin ≥ 8 g/dL
* Serum blood chemistries within 21 days before the first day of radiation, as defined below:

  * Creatinine ≤ 2.0 mg
  * Total bilirubin ≤ 1.5 mg/dL
  * ALT (Alanine Aminotransferase)≤ 3 times the institutional upper limit of normal
  * AST (Aspartate Aminotransferase) ≤ 3 times the institutional upper limit of normal
* Tolerate one text dose (15g) of ascorbate
* Not pregnant
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Recurrent high grade glioma
* G6PD (glucose-6-phosphate dehydrogenase) deficiency
* Patients actively receiving insulin unless approved by the study medical monitor, study sponsor, and the study principal investigator.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide.
* Significant co-morbid central nervous system disease, including but not limited to, multiple sclerosis.
* Patients who are on the following drugs and cannot have a drug substitution: flecainide, methadone, amphetamines, quinidine, and chlorpropamide. High dose ascorbic acid may affect urine acidification and, as a result, may affect clearance rates of these drugs.
* Prior invasive malignancies (except non-melanomatous skin cancers and carcinoma in situ of the cervix or bladder) unless disease free for ≥ 5 years.
* Patients who have received prior chemotherapy (including Gliadel wafers) for the current glioma.
* Prior radiation therapy to the head or neck, which would result in overlap of radiation therapy fields.
* Patients may not be receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because ionizing radiation is a known teratogen, and temozolomide is a Class D agent with the potential for teratogenic or abortifacient effects.
* Known HIV-positive individuals. High-dose ascorbate acid is a known CYP450 3A4 (an enzyme pathway) inducer, which results in lower serum levels of antiretroviral drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Number of grade 3, 4, & 5 adverse events | Weekly during therapy for up to 10 months
  Assess grade 3 and higher adverse events. Evaluate the frequency and severity against the published literature to determine the likely causality between ascorbate and the adverse event(s).

SECONDARY OUTCOMES:
Time to progression | monthly up to 5 years post treatment
  Time from the start of therapy (day 1, cycle 1) to documented disease progression in MRI imaging as described by MacDonald and colleagues.
Overall survival | Up to 5 years
  From start of treatment (cycle 1, day 1) until the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: John M. Buatti, MD, Principal Investigator — Department of Radiation Oncology, The University of Iowa; Joseph J Cullen, MD, Study Director — Professor of Surgery, The University of Iowa
Locations (1):
- Holden Comprehensive Cancer Center at the University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data is shared through an NIH/NCI approved data sharing plan in compliance with subject's consent to sharing. Investigators interested in IPD should contact the sponsor, study PI, or study coordinator for more information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP, and ICF will be shared at conclusion of the study.
Access Criteria: Investigators interested in IPD should contact the sponsor, study PI, or study coordinator for more information. IRB approval for the recipient investigator may be required, as determined by the individual data received.

REFERENCES:
- [Background] Du J, Cullen JJ, Buettner GR. Ascorbic acid: chemistry, biology and the treatment of cancer. Biochim Biophys Acta. 2012 Dec;1826(2):443-57. doi: 10.1016/j.bbcan.2012.06.003. Epub 2012 Jun 20. PMID 22728050
- [Background] Du J, Martin SM, Levine M, Wagner BA, Buettner GR, Wang SH, Taghiyev AF, Du C, Knudson CM, Cullen JJ. Mechanisms of ascorbate-induced cytotoxicity in pancreatic cancer. Clin Cancer Res. 2010 Jan 15;16(2):509-20. doi: 10.1158/1078-0432.CCR-09-1713. Epub 2010 Jan 12. PMID 20068072
- [Result] Schoenfeld JD, Sibenaller ZA, Mapuskar KA, Wagner BA, Cramer-Morales KL, Furqan M, Sandhu S, Carlisle TL, Smith MC, Abu Hejleh T, Berg DJ, Zhang J, Keech J, Parekh KR, Bhatia S, Monga V, Bodeker KL, Ahmann L, Vollstedt S, Brown H, Shanahan Kauffman EP, Schall ME, Hohl RJ, Clamon GH, Greenlee JD, Howard MA, Schultz MK, Smith BJ, Riley DP, Domann FE, Cullen JJ, Buettner GR, Buatti JM, Spitz DR, Allen BG. O2⋅- and H2O2-Mediated Disruption of Fe Metabolism Causes the Differential Susceptibility of NSCLC and GBM Cancer Cells to Pharmacological Ascorbate. Cancer Cell. 2017 Apr 10;31(4):487-500.e8. doi: 10.1016/j.ccell.2017.02.018. Epub 2017 Mar 30. PMID 28366679